CLINICAL TRIAL: NCT07112482
Title: Assessing Cachexia Status in Pakistani Cancer Patients Using the Mini-CASCO Score
Brief Title: Effect of Dietary Counseling and Nutritional Monitoring in Reducing Cancer-related Cachexia Among Female Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Society of Pediatric Oncology (Other)
Collaborators: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Junaid Jamshed, Clinical Research Coordinator, Pakistan Society of Pediatric Oncology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 794/RC/FFH/RWP
Record Dates: First submitted 2025-07-16; First posted 2025-08-08 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Cachexia
Keywords: Cancer-associated cachexia; Randomize Controlled Trail; Dietary Counselling; Nutritional Monitoring; Breast cancer
MeSH Terms: conditions — Breast Neoplasms; Cachexia

STUDY DESIGN:
Intervention Model Description: The intervention group will receive standard oncological care along with tailored dietary counseling and monthly nutritional monitoring for six months. Plans will target 25-30 kcal/kg/day and 1.2-1.5 g/kg/day protein intake, adapted to clinical condition, treatment tolerance, and preferences. Counseling sessions (every 15-21 days) will last 25-30 minutes and address dietary challenges, food tolerance, and symptom-related barriers. Dietary adherence will be tracked using structured food logs and checklists. Light physical activity and psychosocial support will be encouraged. Adherence will be defined as ≥75% session attendance and ≥80% dietary goal achievement.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Oncological Care + Tailored Dietary Counseling + Nutritional Monitoring (Experimental): Participants in the intervention group will receive:
  Standard oncological care (including chemotherapy and other routine cancer treatments) plus
  Individualized dietary counseling: Tailored nutrition plans developed by a clinical dietitian based on energy (25-30 kcal/kg/day) and protein (1.2-1.5 g/kg/day) needs, adjusted for clinical status, dietary tolerance, and treatment side effects.
  Regular nutritional monitoring: Counseling sessions every 15-21 days over a period of six months.
  Dietary adherence tracking: Using structured food records and goal adherence checklists.
  Light physical activity guidance: Encouragement to engage in low-intensity activity appropriate to patient capacity.
  Psychosocial support: Sessions with a certified clinical psychologist to address emotional distress, fatigue, and anorexia.
  Adherence criteria: Defined as attending ≥75% of sessions and meeting ≥80% of dietary goals.
  Interventions: Behavioral: Standard Oncological Care + Tailored Dietary Counseling + Nutritional Monitoring
- Standard Oncological Care (Active Comparator): Participants in this group will receive standard oncological care only, including chemotherapy and other routine cancer treatments, without additional dietary or psychosocial interventions.
  Interventions: Behavioral: Standard Oncological Care + Tailored Dietary Counseling + Nutritional Monitoring

INTERVENTIONS:
Behavioral: Standard Oncological Care + Tailored Dietary Counseling + Nutritional Monitoring — Participants in this group will receive:
  Standard oncological care (e.g., chemotherapy and routine cancer treatments)
  Individualized dietary counseling: Nutrition plans tailored by a clinical dietitian to meet energy needs (25-30 kcal/kg/day) and protein needs (1.2-1.5 g/kg/day), adapted to clinical status, dietary tolerance, and treatment side effects.
  Regular nutritional monitoring: Counseling sessions every 15-21 days over a period of six months.
  Dietary adherence tracking: Through structured food records and goal adherence checklists.
  Light physical activity guidance: Encouragement to engage in low-intensity activity suited to patient capacity.
  Psychosocial support: Sessions with a certified clinical psychologist addressing emotional distress, fatigue, and anorexia.
  Adherence criteria: Defined as attending ≥75% of sessions and meeting ≥80% of dietary goals.

SUMMARY:
In this parallel, two-arm randomized controlled trial (RCT), 140 female patients with advanced-stage breast cancer and clinical features of cachexia will be randomized using block-stratified allocation into an intervention group (n = 70) and a control group (n = 70). The intervention group will receive standard oncological care along with personalized dietary counseling and monthly nutritional monitoring for six months, whereas the control group will receive standard care alone. The severity of cachexia will be assessed at baseline and follow-up using the Mini-CASCO tool, which will evaluate five domains: body composition, inflammatory-metabolic profile (C-reactive protein, serum albumin, hemoglobin, absolute lymphocyte count), physical performance (Eastern Cooperative Oncology Group [ECOG] status), anorexia (Simplified Nutritional Appetite Questionnaire [SNAQ]), and quality of life (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 [EORTC QLQ-C30]).

DETAILED DESCRIPTION:
This randomized controlled trial evaluates the impact of individualized dietary counseling with ongoing nutritional monitoring on cancer cachexia severity in women with advanced breast cancer. Cancer cachexia is a multifactorial syndrome characterized by muscle wasting, anorexia, inflammation, and reduced functional status, significantly impairing quality of life and treatment tolerance. Despite its clinical relevance, targeted interventions for cachexia remain underutilized in routine oncology care.

The study is designed as a two-arm, parallel-group trial comparing standard oncological care alone with standard care plus a tailored nutritional intervention. The intervention is structured to address energy and protein intake requirements using individualized plans developed by a clinical dietitian. It incorporates scheduled nutritional counseling sessions, structured adherence monitoring through food logs and checklists, and reinforcement strategies including light physical activity promotion and psychosocial support.

To ensure methodological rigor, the study employs block-stratified randomization with concealed allocation using opaque, sealed envelopes. While blinding of participants and care providers is not feasible due to the nature of the intervention, outcome assessors and data analysts will be blinded to minimize bias. The primary outcome-change in cachexia severity over six months-will be evaluated using a validated multidimensional tool that captures clinical, functional, and patient-reported parameters.

Data will be entered into a secure, password-protected database with built-in quality control processes, including double data entry and discrepancy checks. Missing data will be handled using multiple imputation under the assumption of missing at random. Statistical analyses will be conducted on an intention-to-treat basis, with appropriate covariate adjustment and effect size reporting.

This trial is expected to provide practical evidence on the feasibility and effectiveness of structured, individualized nutritional interventions as part of supportive oncology care in resource-constrained settings.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 20 to 60 years
2. Histologically confirmed advanced breast cancer
3. Documented unintentional weight loss of ≥5% over the past 6 months
4. Hemoglobin level <12 g/dL or average daily energy intake <1500 kcal/day
5. Ability to provide written and verbal informed consent

Exclusion Criteria:

1. Malnutrition due to non-cancer causes (e.g., chronic starvation, eating disorders)
2. Presence of chronic gastrointestinal or endocrine disorders affecting nutritional status (e.g., Crohn's disease, Cushing's syndrome)
3. Current pregnancy or lactation
4. Concurrent diagnosis of another malignancy
5. Any condition that, in the opinion of the investigator, may interfere with study participation or outcomes (e.g., severe psychiatric illness, cognitive impairment)

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Change in cachexia severity measured by the Mini-CASCO composite score | From baseline to 6 months
  The primary outcome will be the change in cachexia severity from baseline to six months, measured using Mini-CASCO, which includes:
  Body Composition (40%): Body weight and lean body mass assessed by digital scale and BIA.
  Inflammatory/Metabolic/Immune Status (20%): CRP, albumin, hemoglobin, and lymphocyte count.
  Physical Performance (15%): ECOG scale, handgrip strength, stair climbing, and fatigue assessments.
  Anorexia (15%): SNAQ scores, 24-hour recall, and food frequency questionnaires.
  The Mini-Cancer Cachexia Score (Mini-CASCO) is a validated multidimensional scoring system that assesses cancer cachexia severity using five domains: body composition, inflammation/metabolism, physical performance, anorexia, and quality of life. The total score ranges from 0 to 100, with higher scores indicating more severe cachexia.

SECONDARY OUTCOMES:
Change in Body Weight | From baseline to 6 months
  Change in body weight measured using a calibrated digital scale.
Change in Lean Body Mass | From baseline to 6 months
  Kilograms (kg) Description: Change in lean mass assessed via Bioelectrical Impedance Analysis (BIA).
Change in C-Reactive Protein (CRP) | From baseline to 6 months
  Description: Assessed as a marker of systemic inflammation. Milligrams per liter (mg/L)
Change in ECOG Performance Status | From baseline to 6 months
  Eastern Cooperative Oncology Group (ECOG) performance score; higher values indicate worse performance. ECOG scale (0-5)
Change in SNAQ Score (Simplified Nutritional Appetite Questionnaire) | From baseline to 6 months
  Lower scores indicate higher risk of weight loss. SNAQ score (4-20)
Change in Quality of Life (EORTC QLQ-C30, Urdu version) | From baseline to 6 months
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ-C30), global health status scale; higher scores indicate better quality of life. Global Health Status/QoL scale (0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Research Coordinator, MSPH, DrPH, Study Chair — Pakistan Institute of Medical Sciences
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Yes, individual participant data (IPD) will be shared. The following data will be shared: de-identified demographic data, baseline characteristics, outcome data, and adverse events. Data will be available beginning 6 months after publication and will be shared for a period of 3 years. Data will be accessible to researchers with a methodologically sound proposal via a secure data-sharing platform, upon request to the principal investigator.
Supporting Information: Study Protocol
Time Frame: IPD will be available starting 6 months after publication of the primary results and will remain accessible for 3 years.
Access Criteria: IPD will be available to researchers with a methodologically sound proposal. Requests must be submitted in writing to the principal investigator and must include a study protocol and ethical approval. Data will be provided through a secure data access system upon signing a data-sharing agreement.

DOCUMENTS (3):
  • Study Protocol (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT07112482/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT07112482/SAP_001.pdf
  • Informed Consent Form (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT07112482/ICF_002.pdf